CLINICAL TRIAL: NCT02615587
Title: Burden of Illness in Atrial Fibrillation in Denmark
Brief Title: Burden of Illness in Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18313
Record Dates: First submitted 2015-10-07; First posted 2015-11-26 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Atrial Fibrillation
Keywords: non-valvular Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AF patients in Denmark / Cohort 1: The base population of AF patients for diagnosis and health care utilization / resource use will be identified in the National Patient Registry. For a given period of time (2000-2013, both years inclusive) all patients with a hospital contact (admission, outpatient visit or ER visit) and for whom AF was the primary or secondary diagnosis code will be identified.
  Further Data sources used:
  Registry of Medicinal Product Statistics: for determining the individuals' use of prescription medicine DREAM database: for investigation of sickness benefit and productivity loss Statistics Denmark's databases: on social services from municipalities Cause of Death Registry: AF-patients or controls who died during the study period (2000-2013) Danish Civil Registry: used for identification of controls, holds information about age, gender
  Interventions: Drug: Standard of care in AF in Denmark

INTERVENTIONS:
Drug: Standard of care in AF in Denmark — As used in clinical practice, analysed as per drug class, not separate drugs.

SUMMARY:
The overall goal of this retrospective registry study is to investigate the burden-of.illness in atrial fibrillation (AF) in Denmark. Several Danish registries will be utilized to collect information on the diseases epidemiology including incidence and prevalence of AF and stroke as well as a stroke risk stratification of the Danish AF-population, the clinical and economical burden (in terms of direct and indirect cost) of AF and stroke to Danish patients, healthcare providers / healthcare system and society as well as describing treatment patterns with anticoagulant agents and their consequences in terms of stroke, bleeds, death and according cost in a real-life setting.

ELIGIBILITY:
Inclusion Criteria:

* Primary and secondary diagnosis with AF;
* The base population of AF patients will be identified in the National Patient Registry. For a given period of time (2000-2013, both years inclusive) all patients with a hospital contact (admission, outpatient visit or ER visit) and for whom AF was the primary or secondary diagnosis code (ICD10-code: DI480, DI481, DI482, DI483, DI484, DI489) will be included.

Exclusion Criteria:

* Patients younger than 18 and older than 90 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The base population of AF patients will be identified in the National Patient Registry. For a given period of time (2000-2013, both years inclusive) all patients with a hospital contact (admission, outpatient visit or ER visit) and for whom AF was the primary or secondary diagnosis code will be identified.
Sampling Method: Non-Probability Sample
Enrollment: 107532 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with (non-valvular) AF in total Danish population and by gender and age groups 18-65, 66-75, 75+, 80+ | up to 4 weeks
Number of newly diagnosed patients with (non-valvular) AF per year in total Danish population and by gender and age groups 18-65, 66-75, 75+, 80+ | up to 4 weeks
Number of patients with (non-valvular) AF per Danish Region and by gender and age groups 18-65, 66-75, 75+, 80+ | up to 4 weeks
Number of newly diagnosed patients with (non-valvular) AF per year and per Danish Region and by gender and age groups 18-65, 66-75, 75+, 80+ | up to 4 weeks
Mortality among AF patients compared with that of the general population/the 'controls', if possible by gender and age group | up to 4 weeks
Number of patients with stroke in (non-valvular) AF-patients in Denmark by gender and age groups 18-65, 66-75, 75+, 80+ | up to 4 weeks
Number of newly diagnosed patients with stroke in (non-valvular) AF-patients per year in Denmark by gender and age groups 18-65, 66-75, 75+, 80+ | up to 4 weeks
Mortality among stroke patients (in AF) compared with that of the population/the 'controls' and the total AF-population, if possible by gender and age group | up to 4 weeks
Direct cost in AF (in total and per patient) | up to 4 weeks
  Costs due to:
  Patients' resource use in the primary care sector (GP-visits, etc.) Patients' resource use in the hospital sector, including specialized rehabilitation Patients' use of prescription medicine
  Cost will be shown:
  For Denmark Per Region including differences between Regions For differentiation by age group For differentiation by Region and age group, if possible based on sample sizes
Direct cost in AF-related stroke (in total and per patient) | up to 4 weeks
  Costs due to:
  Patients' resource use in the primary care sector (GP-visits, etc.) Patients' resource use in the hospital sector, including specialized rehabilitation Patients' use of prescription medicine
  Cost will be shown:
  For Denmark Per Region including differences between Regions For differentiation by age group For differentiation by Region and age group, if possible based on sample sizes
Indirect cost in AF (in total and per patient) | up to 4 weeks
  Costs due to:
  Patients' long-term absence from the labour force (only relevant for patients under 65 years of age) Patients' demand for home care and rehabilitation delivered by municipalities
  Cost will be shown:
  For Denmark Per Region including differences between Regions For differentiation by age group For differentiation by Region and age group, if possible based on sample sizes
Indirect cost in AF-related stroke (in total and per patient) | up to 4 weeks
  Costs due to:
  Patients' long-term absence from the labour force (only relevant for patients under 65 years of age) Patients' demand for home care and rehabilitation delivered by municipalities
  Cost will be shown:
  For Denmark Per Region including differences between Regions For differentiation by age group For differentiation by Region and age group, if possible based on sample sizes

SECONDARY OUTCOMES:
Number of patients with AF-related stroke rated per CHADS2-score (0 to 6) in Danish population | up to 4 weeks
  CHADS2-score: Congestive heart failure/left ventricular dysfunction, Hypertension, Age, Diabetes, Stroke (Doubled)
Percentage (%) of patients with AF-related stroke rated per CHADS2-score (0 to 6) in Danish population | up to 4 weeks
  CHADS2-score: Congestive heart failure/left ventricular dysfunction, Hypertension, Age, Diabetes, Stroke (Doubled)
Number of patients with AF-related stroke rated per average CHADS-score in Danish population | up to 4 weeks
Percentage (%) of patients with AF-related stroke rated per average CHADS-score in Danish populationPercentage (%) of patients with AF-related stroke rated per average CHADS-score in Danish population | up to 4 weeks
Number of patients with AF-related stroke rated per CH2ADS2-VASc-score (0 to 9) in Danish population | up to 4 weeks
Percentage (%) of patients with AF-related stroke rated per CH2ADS2-VASc-score (0 to 9) in Danish population | up to 4 weeks
Number of patients per HAS-BLED-score (0 to 9) in Danish AF-population | up to 4 weeks
Percentage (%) of patients per HAS-BLED-score (0 to 9) in Danish AF-population | up to 4 weeks
Number of patients per average HAS-BLED-score in Danish AF-population | up to 4 weeks
Percentage (%) of patients per average HAS-BLED-score in Danish AF-population | up to 4 weeks
Number of patients in total and per CH2ADS2-VASc-score receiving Acetylsalicylic Acid [ASA] | up to 4 weeks
Number of patients in total and per CH2ADS2-VASc-score receiving warfarin | up to 4 weeks
Number of patients in total and per CH2ADS2-VASc-score receiving any Novel Oral Anticoagulants [NOACs] | up to 4 weeks
Number of patients in total and per CH2ADS2-VASc-score receiving no treatment | up to 4 weeks
Percentage (%) of patients in total and per CH2ADS2-VASc-score receiving Acetylsalicylic Acid [ASA] | up to 4 weeks
Percentage (%) of patients in total and per CH2ADS2-VASc-score receiving Warfarin | up to 4 weeks
Percentage (%) of patients in total and per CH2ADS2-VASc-score receiving any Novel Oral Anticoagulants [NOACs] | up to 4 weeks
Percentage (%) of patients in total and per CH2ADS2-VASc-score receiving no treatment | up to 4 weeks
Number of patients experiencing events (e.g. stroke, Systemic Embolism [SE], Myocardial Infarction [MI], bleeds, death) since AF-diagnosis per anticoagulant agent (AC)-medication incl. no treatment in total | up to 4 weeks
Percentage (%) of patients experiencing events (e.g. stroke, Systemic Embolism [SE], Myocardial Infarction [MI], bleeds, death) since AF-diagnosis per anticoagulant agent (AC)-medication incl. no treatment in total | up to 4 weeks
Number of patients experiencing events (e.g. stroke, Systemic Embolism [SE], Myocardial Infarction [MI], bleeds, death) since AF-diagnosis per Anticoagulant agent (AC)-medication incl. no treatment per CHADS-VASc-score | up to 4 weeks
Percentage (%) of patients experiencing events (e.g. stroke, Systemic Embolism [SE], Myocardial Infarction [MI], bleeds, death) since AF-diagnosis per Anticoagulant agent (AC)-medication incl. no treatment per CHADS-VASc-score | up to 4 weeks
Vitamin K antagonist (VKA) treated AF-patients in AC-clinics versus GP-setting | up to 4 weeks
  Based on data from the National Patient Registry, the Primary Care Registry and the Registry of Medicinal Product Statistics and inclusion codes for specific fees/services, it will be possible to identify which patients are treated in an AC-clinic and which patients are treated in a GP-setting
Direct and indirect cost of AC medication treatment patterns | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Denmark